CLINICAL TRIAL: NCT07181551
Title: Forward to Quit: A Person-centered Mobile Technology Intervention for Smoking Cessation Among Transgender Adults
Acronym: F2Q
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-2296; 5R34DA058191-03 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F2Q Intervention (Experimental): Participants will receive access to the Forward to Quit (F2Q) mHealth smoking cessation intervention tailored for transgender adults
  Interventions: Behavioral: Forward to Quit (F2Q)

INTERVENTIONS:
Behavioral: Forward to Quit (F2Q) — A mobile health (mHealth) smoking cessation intervention designed specifically for transgender adults. Delivered via a secure website accessible by smartphone or tablet.

SUMMARY:
This study evaluates the feasibility, acceptability, and preliminary efficacy of "Forward to Quit" (F2Q), a person-centered mobile health (mHealth) smoking cessation intervention designed specifically for transgender adults. The intervention was developed in collaboration with transgender individuals and gender-affirming healthcare providers. The study includes usability testing and a remote single-arm pilot trial. Primary outcomes include feasibility and acceptability of both the intervention and remote biochemical verification of smoking cessation. Secondary outcomes include self-reported and biochemically verified smoking cessation, as well as changes in psychosocial factors such as social support and gender affirmation. The goal is to inform a future large-scale trial and address tobacco-related health disparities in transgender populations.

ELIGIBILITY:
Inclusion Criteria:

* Identify with a gender different from sex assigned at birth
* 18+ years of age
* Report smoking at least 5 cigarettes per day
* Have smoked 100+ cigarettes in their lifetime
* Own a device that can access the Internet (e.g., tablet, smartphone)
* Speak English
* Be willing to submit biochemical samples to verify cessation
* Be willing to use a website-based intervention to help with quit attempt
* Be willing to set a quit date within 1 month of baseline assessment
* Be willing to complete 3 months post-baseline and 6 months post-baseline assessments

Exclusion Criteria:

* Do not meet inclusion criteria
* Medical conditions precluding use of the carbon monoxide (CO) monitor or salivary cotinine testing
* Current use of pharmacotherapies for nicotine dependence
* Enrollment in another tobacco cessation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability | 3 months post-baseline
  We will assess participants' perceptions of information quality and usefulness as well as overall satisfaction with the intervention. If the average score across all items is >=6 on a 7-point scale for 90% of participants after using intervention for 3 months, we will consider intervention to be acceptable.
Intervention feasibility | 3 months post-baseline
  Feasibility will be met if retention rates are at least 80%.
Remote biochemical data collection acceptability | 3 month post-baseline
  We will measure participants' perceived difficulty, satisfaction, and comfort with remote biochemical verification. If scores are >=6 on a 7-point scale for 90% of participants, we will consider remote biochemical verification to be acceptable.
Remote biochemical data collection feasibility | 3 months post-baseline
  Completion rate (percentage of eligible participants who submit biochemical samples for verification of tobacco abstinence)

SECONDARY OUTCOMES:
Smoking cessation | 3 month post-baseline
  Participants will be categorized as abstinent or not abstinent based on self-report.
Conceptual model covariates | 3 months post-baseline
  Nicotine dependence and other conceptual model covariates will be assessed with validated survey items.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Sun, PhD, Principal Investigator — Universtiy of Colorado Anschutz Medical Campus

IPD SHARING:
Plan to Share IPD: Undecided
Unsure of where or how IPD would be shared